CLINICAL TRIAL: NCT01899352
Title: Procedures, Complications and Follow-up of Tracheostomy in Intensive Care Units - a Prospective Study by Italian Society of Anesthesia, Analgesia, Resuscitation and Intensive Care (SIAARTI)
Brief Title: Procedures, Complications and Follow-up of Tracheostomy in Intensive Care Units.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Genova (Other)
Responsible Party: Principal Investigator, Paolo Pelosi, Professor-head of intensive care unit, University of Genova
Allocation: Non-Randomized | Model: Single Group | Masking: Single
Other Study IDs: PCF-TracheoTrial
Record Dates: First submitted 2013-07-02; First posted 2013-07-15 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Respiratory Failure; Neurological Disease; Heart Failure; Airway Management
MeSH Terms: conditions — Respiratory Insufficiency; Nervous System Diseases; Heart Failure | interventions — Tracheostomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tracheostomy (Other): The investigators will enroll all the critical ill patients undergoing tracheostomy performed in intensive care units
  Interventions: Procedure: Tracheostomy

INTERVENTIONS:
Procedure: Tracheostomy — Percutaneous and surgical tracheostomies will be performed with the procedure currently available in clinical practice.

SUMMARY:
Tracheostomy is worldwide used for critically ill patients. The aim of our study is to assess the mortality, quality of life, laryngeal function, procedures, early and late complications of tracheostomy performed for critically ill patients admitted in intensive care units.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* indications for tracheostomy

Exclusion Criteria:

* Infection/inflammation of neck tissue
* Previous neck surgery causing abnormal anatomy of the site
* Recent surgery of cervical spine

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Mortality at ICU discharge | within 2 days after discharge

SECONDARY OUTCOMES:
Quality of Life | within 2 days after discharge, at 3, 6 and 12 months after tracheostomy
  Quality of life will be evaluated at 3, 6 and 12 months after the discharge from the intensive care unit.
Laryngeal organ function | within 2 days after discharge, at 3, 6 and 12 months after tracheostomy
  Laryngeal organ function will be evaluated at 3, 6 and 12 months after the discharge from intensive care unit.
Late complications | from day 2 until the discharge
Procedural findings of percutaneous tracheostomy | at the beginning and at the end of tracheostomy procedures
Early complication | in the first 24 hours from the end of the procedure

CONTACTS AND LOCATIONS:
Locations (10):
- Italy (10):
  - Italian Society of Anesthesia, Analgesia, Resuscitation and Intensive Care, Assisi, Italy
  - Policlinico Vittoio Emanuele, Catania, Italy
  - Policlinico SS Annunziata, Chieti, Italy
  - Intensive care unit - San Martino-IST, Genoa, Italy
  - IRCCS Azienda Ospedaliera San Martino IST, Genoa, Italy
  - Centro Cardiologico Monzino, Milan, Italy
  - University of Naples "Federico II", Naples, Italy
  - Ospedale Morgagni-Pierantoni, Rimini, Italy
  - Università Cattolica del Sacro Cuore, Rome, Italy
  - Università di Torino, Turin, Italy

REFERENCES:
- [Derived] Vargas M, Battaglini D, Antonelli M, Corso R, Frova G, Merli G, Petrini F, Ranieri MV, Sorbello M, Di Giacinto I, Terragni P, Brunetti I, Servillo G, Pelosi P. Follow-up short and long-term mortalities of tracheostomized critically ill patients in an Italian multi-center observational study. Sci Rep. 2024 Jan 28;14(1):2319. doi: 10.1038/s41598-024-52785-y. PMID 38281994